CLINICAL TRIAL: NCT07145437
Title: Evaluation of the Prognostic Value of Radio-induced Lymphocyte Apoptosis for Predicting Late Radiation-induced Toxicities After Stereotactic Body Radiotherapy in Patients With Localized Prostate Cancer
Brief Title: Prostate Stereotactic Radiation and Radio-induced Lymphocyte Apoptosis for Predicting Late Toxicities in Prostate Cancer (PROSTERA)
Acronym: PROSTERA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Sainte Clotilde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A00340-49
Record Dates: First submitted 2025-08-11; First posted 2025-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Stereotactic Body Radiotherapy; Late Toxicity; RILA; Predictive Biomarker; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: SBRT + RILA assay (single-arm) (Experimental): All participants assigned to this single experimental arm will receive stereotactic body radiotherapy (SBRT) to the prostate delivered according to the PROSTERA protocol with predefined dose prescription and organ-at-risk constraints. A single peripheral blood sample (2 mL, lithium-heparin) will be collected at the time of CT simulation for the Radio-induced Lymphocyte Apoptosis (RILA) assay. Samples are transported and processed at the designated laboratory (LIRS) and handled per the RILA SOP: processing within 4 hours of collection, incubation 16-24 hours, ex-vivo irradiation (8 Gy), further incubation 48 hours, staining for CD4/CD8 and propidium iodide, and flow cytometry analysis (10,000 events, measured in triplicate) to quantify apoptotic T-lymphocytes. RILA results will be used for correlative and prognostic analyses versus late genitourinary and gastrointestinal toxicities (CTCAE v5.0), PSA kinetics and patient-reported outcomes (EORTC QLQ-PR25, QLQ-C30, IPSS).
  Interventions: Diagnostic Test: Radio-induced Lymphocyte Apoptosis (RILA) Assay; Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Diagnostic Test: Radio-induced Lymphocyte Apoptosis (RILA) Assay — peripheral blood sample processed via the RILA assay to quantify apoptotic CD8+/CD4+ T cells following ex vivo irradiation.
Radiation: Stereotactic body radiotherapy (SBRT) — SBRT delivered to the prostate with image guidance, respecting dose constraints for organs at risk;

SUMMARY:
This monocentric interventional study investigates whether the Radio-induced Lymphocyte Apoptosis (RILA) assay can predict the occurrence of late radiation-induced toxicities in patients with localized prostate cancer treated with stereotactic body radiotherapy (SBRT). Eligible patients will undergo a peripheral blood sample collection for the RILA test prior to SBRT. Toxicities will be assessed using CTCAE v5.0 criteria, and quality of life will be evaluated with EORTC QLQ-PR25, QLQ-C30, and IPSS questionnaires over a 60-month follow-up. The results aim to optimize patient selection for SBRT and reduce the risk of severe late side effects.

DETAILED DESCRIPTION:
PROSTERA is a prospective, single-arm, monocentric interventional study (RIPH-2) designed to evaluate the prognostic performance of the Radio-induced Lymphocyte Apoptosis (RILA) assay to predict late radiation-induced toxicities in patients with localized prostate cancer treated with stereotactic body radiotherapy (SBRT).

The primary objective is to determine whether pre-treatment RILA (percentage of apoptotic T-lymphocytes measured ex-vivo after controlled irradiation) is predictive of clinically meaningful late toxicities graded ≥2 according to CTCAE v5.0 within 24 months after SBRT. Secondary objectives include PSA kinetics, patient-reported outcomes (EORTC QLQ-PR25, QLQ-C30 and IPSS), dosimetric correlations, and estimation of diagnostic performance metrics (AUC, sensitivity, specificity) of the RILA assay.

A single peripheral blood sample (2 mL) is collected at the time of CT simulation (inclusion visit). Samples are transported to the designated laboratory (LIRS/RunResearch) and processed according to the RILA SOP: cells are placed in culture (RPMI 1640 + 20% FBS, dilution 1:10) within 4 hours of collection, incubated 16-24 hours, then irradiated ex-vivo (8 Gy; conformational irradiation using institutional accelerator) and incubated for an additional 48 hours. After post-irradiation incubation cells are stained for CD4/CD8 and propidium iodide and analysed by flow cytometry (FACS) on 10,000 events in triplicate to derive the percentage of apoptotic CD4+ and CD8+ T-cells. All assay timings and plate/aliquot identifiers are recorded in laboratory logs. The collected sample is entirely consumed for the assay (no sample retention).

Eligible participants are adult males with localized prostate adenocarcinoma meeting the protocol inclusion criteria (e.g. clinical stage T1-T2, Gleason score 6-7, PSA <15 ng/mL as per protocol), able to provide written informed consent and compliant with follow-up procedures. Key exclusions include prior pelvic radiotherapy, metastatic disease, inability to consent, and other criteria listed in the protocol. Enrollment will be consecutive to limit selection bias.

All participants receive SBRT delivered according to institutional conformational technique (protocol-specified dose constraints and organ-at-risk delineation per RTOG recommendations; typical stereotactic schedule described in the protocol). Imaging data (centering CT and any low-dose CT), treatment plans and dose-volume histograms (DVH) will be collected and stored in the electronic CRF for dose-toxicity correlation analyses.

Safety and patient-reported outcomes will be recorded during routine follow-up visits at baseline (pre-SBRT) and at 1, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months post-radiotherapy; CTCAE v5.0 will be used for toxicity grading and the EORTC QLQ-PR25, QLQ-C30 and IPSS questionnaires for quality-of-life and urinary symptom assessment. PSA will be measured at the same scheduled timepoints. No additional study-specific clinic visits are required beyond standard care.

The planned sample size is 220 subjects (calculated to achieve the desired precision for the RILA AUC estimate; ~166 evaluable subjects minimally required), with an anticipated inclusion period of 24 months and maximum individual follow-up of 61 months (total study duration ≈ 88 months). Data will be recorded in a pseudonymized electronic CRF and source documents will remain available in patient medical records. The study will be conducted under the applicable ethical and regulatory framework (CPP approval, MR-001, GDPR).

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 60 years or older, presenting with localized prostate cancer of low or intermediate risk (T1-T2 stage, Gleason score 6-7, and PSA <15 ng/mL) without metastatic disease, and for whom radiotherapy is indicated.
* Patient affiliated with, or beneficiary of, the French national health insurance system.
* French-speaking patient.
* Patient who has been informed about the study and has provided written informed consent.

Exclusion Criteria:

* Patient unable to read, write, or understand French.
* Vulnerable patient as defined in Article L1121-6 of the French Public Health Code.
* Adult under legal guardianship, curatorship, or judicial protection.
* Patient unable to personally provide informed consent as per Article L1121-8 of the French Public Health Code, or adult protected by law.
* Patient already enrolled in an interventional study that could influence the outcomes of the present study.
* Patient with a history of prostate and/or digestive surgery.
* Refusal to sign the written informed consent at inclusion.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male patients with localized prostate cancer
Enrollment: 220 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of one or more late radiation-induced complications | 24 months post-stereotactic radiotherapy
  Number of participants presenting one or more late radiation-induced complications, assessed using the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

SECONDARY OUTCOMES:
Mortality rate of T-CD8+/-CD4+ lymphocytes | After in vitro culture and irradiation at 8 Gy
  Percentage of T-CD8+/-CD4+ lymphocytes mortality measured by flow cytometry after in vitro culture of blood samples and irradiation at 8 Gy.
Clinical and biological variables of patients | At baseline and during follow-up (up to 60 months post-radiotherapy)
  Evaluation of clinical and biological variables (e.g., blood counts, PSA, comorbidities) collected during follow-up.
  Unit of Measure: Values according to each variable (e.g., PSA ng/mL, blood counts G/L, yes/no for comorbidities)
Quality of life - EORTC QLQ-PR25 | Baseline, 1, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months post-radiotherapy
  Scores reported according to the validated scale (0-100). Higher scores = worse symptoms/problems, better functioning for functional scales.
  Score (0-100)
Quality of life - EORTC QLQ-C30 | Baseline, 1, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months post-radiotherapy
  Scores reported according to the validated scale (0-100). Higher scores = worse symptoms, better functioning for functional/global health. Unit of Measure: Score (0-100)
Urinary symptoms - International Prostate Symptom Score (IPSS) | Baseline, 1, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months post-radiotherapy
  Validated 0-35 scale, where higher scores = worse urinary symptoms. Unit of Measure: Score (0-35)
Treatment tolerance - Number of participants with adverse events | Baseline, 1, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months post-radiotherapy
  Graded according to CTCAE v5.0 (Grades 1-5).

CONTACTS AND LOCATIONS:
Overall Officials: Mickael DR Begue, Doctor, Principal Investigator — Clinique Sainte Clotilde

IPD SHARING:
Plan to Share IPD: Undecided